CLINICAL TRIAL: NCT00876590
Title: Glucose Monitor Accuracy Investigation (Ⅱ)
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Feng-Huei Lin, Biomedical Engineering Department of National Taiwan University Hospital
Other Study IDs: 9461701248
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
According to Section 7.3 and Section 7.4, ISO 15197(2003), it adopts the whole blood of fingertips as samples to evaluate the accuracy of portable BGM.

DETAILED DESCRIPTION:
The clinical medical technologists collected blood samples from 319 volunteers including 90 diabetics and 229 healthy people. The range of the blood glucose concentration was from 30.2mg/dL to 577.5mg/dL. The result of clinic evaluation shows that the accuracy of BGM matches the requirement of ISO15197(2003).

ELIGIBILITY:
Inclusion Criteria:

* volunteers with diabetes and non-diabets

Exclusion Criteria:

* hypertension,fever,AIDS,hemophilia

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The glucose concentrations of volunteer shall be distributed as specified in ISO15197 Table 3
Sampling Method: Non-Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2006-04; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
glucose | 10 min

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Huei Lin, PhD, Study Director — Biomedical Engineering Department of National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan